CLINICAL TRIAL: NCT04065347
Title: Quantification of Tenofovir Alafenamide Adherence and Exposure in Adults Living With HIV
Brief Title: Quantification of Tenofovir Alafenamide Adherence (QUANTI-TAF)
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-0715; 1R01AI145453-01A1 (NIH)
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: HIV/AIDS; Adherence, Medication
Keywords: Adherence; Dried Blood Spots; Tenofovir-diphosphate; Antiretroviral therapy; Tenofovir alafenamide
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: A total of 150 participants taking tenofovir alafenamide will be enrolled in this cohort.
  Interventions: Device: Digital Pill
- Group 2: A total of 30 participants initiating/re-initiating tenofovir alafenamide will be enrolled in this cohort.
  Interventions: Device: Digital Pill

INTERVENTIONS:
Device: Digital Pill — Digital Pill over encapsulating tenofovir alafenamide ART
  Other Names: etectRx ID-Cap System

SUMMARY:
This study is being done to evaluate the relationship between adherence to antiretroviral therapy (ART) and HIV drug concentrations in persons living with HIV (PLWH) that are taking tenofovir alafenamide (TAF). Adherence will be measured with an ingestible biosensor (digital pill). Antiretroviral drug concentrations will be measured in different types of blood cells.

DETAILED DESCRIPTION:
PLWH taking or initiating/re-initiating TAF will be recruited for a 16-week study. Upon entering the study, participants will be trained on the use the digital pill to objectively quantify adherence. Study participants already taking TAF will return every 4 weeks for a study visit where blood for drug concentrations will be obtained. Participants initiating/re-initiating TAF will return weekly for the first 4 weeks, at weeks 6 and 8, and every 4 weeks thereafter for a study visit where drug concentrations will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males with HIV, able to give informed consent and comply with study procedures.
2. Currently on (> 6 months), or planning to initiate/re-initiate TAF.

Exclusion Criteria:

1. For females of childbearing age, active pregnancy or any intent to become pregnant
2. Hepatitis C (HCV) infection for which treatment is anticipated within the next 16 weeks after enrollment. Treated HCV with sustained virologic response is allowable if last dose of HCV antivirals was >12 months prior to enrollment
3. Advanced renal (eGFR <30 mL/min/1.73m**2) or liver (Child-Pugh B or C) disease
4. History of extensive bowel surgery, gastric bypass, or gastroparesis
5. Concomitant use of any prescription or non-prescription drug known (or with the potential) to significantly influence the PK of TAF (e.g. rifamycins, carbamazepine, phenytoin, St. John's Wort, tipranavir)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLWH who are initiating/re-initiating or have been on TAF for > 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Tenofovir-diphosphate (TFV-DP) in Dried Blood Spots (DBS) | Week 12
  Steady-state drug concentration distribution and quantiles for highly adherent (i.e. >95% of ingestions) participants.
Tenofovir-diphosphate (TFV-DP) in Dried Blood Spots (DBS) | Week 16
  Steady-state drug concentration distribution and quantiles for highly adherent (i.e. >95% of ingestions) participants.

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Anderson, PharmD, Principal Investigator — University of Colorado-AMC
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coyle RP, Morrow M, Mann SC, Mainella V, Ellis SL, Schwab S, Coppinger C, Barker N, Ellison L, Zheng JH, Al Zuabi S, Alpert PE, Carnes TC, Buffkin DE Jr, Chai PR, Bushman LR, Kiser JJ, MaWhinney S, Brooks KM, Anderson PL, Castillo-Mancilla JR. Tenofovir-Diphosphate and Emtricitabine-Triphosphate Adherence Benchmarks in Dried Blood Spots for Persons With HIV Receiving Tenofovir Alafenamide and Emtricitabine-Based Antiretroviral Therapy (QUANTI-TAF). Clin Infect Dis. 2024 Nov 22;79(5):1233-1241. doi: 10.1093/cid/ciae212. PMID 38636950